CLINICAL TRIAL: NCT00416923
Title: Phase I Study of Intrathecal Rituximab in Patients With Recurrent CNS Lymphoma
Brief Title: Intrathecal Rituximab in Treating Patients With Recurrent CNS Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000454842; UCSF-01302; UCSF-H9414-19588-04; UCSF-U2337S; GENENTECH-UCSF-01302
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Brain and Central Nervous System Tumors; Lymphoma
Keywords: recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; primary central nervous system non-Hodgkin lymphoma; leptomeningeal metastases; intraocular lymphoma; AIDS-related primary CNS lymphoma; Waldenström macroglobulinemia; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Lymphoma; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Meningeal Carcinomatosis; Intraocular Lymphoma; Waldenstrom Macroglobulinemia | interventions — Rituximab

ARMS (1):
- intrathecal rituximab (Experimental): 3 dose levels of intrathecal rituximab, 10mg, 25mg, 50mg
  Interventions: Biological: rituximab

INTERVENTIONS:
Biological: rituximab

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving rituximab intrathecally may be an effective treatment for recurrent CNS lymphoma.

PURPOSE: This phase I trial is studying the side effects and best dose of intrathecal rituximab in treating patients with recurrent CNS lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and pharmacokinetics of intrathecal rituximab in patients with recurrent CNS lymphoma arising from CD20+ B-cell non-Hodgkin's lymphoma.

Secondary

* Determine the efficacy of intrathecal rituximab.
* Determine the molecular pathogenesis of lymphomatous meningitis.
* Determine the molecular basis for response or lack of response to rituximab.
* Identify molecular markers specific for lymphomatous meningitis that will be useful for prognostic evaluation of peripheral lymphomas.
* Determine the quality of life of patients treated with intrathecal rituximab.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive rituximab intrathecally over 10 minutes on day 1 in week 1 and on days 1 and 4 in weeks 2-5 in the absence of disease progression or unacceptable toxicity. Patients achieving at least a partial response with no rituximab-related neurotoxicity may continue to receive treatment beyond 5 weeks.

Cohorts of patients receive escalating doses of rituximab until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which fewer than 1/3 of patients experience dose-limiting toxicity.

Quality of life is assessed at baseline and at the completion of study treatment.

After completion of study treatment, patients are followed periodically for 5 years.

PROJECTED ACCRUAL: A total of 10 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Cytologically confirmed relapsed CNS lymphoma

  * Arising from primary CNS lymphoma or systemic non-Hodgkin's lymphoma
* Evidence of brain parenchymal involvement, cerebrospinal fluid (CSF) involvement, or ocular involvement after radiation treatment or intrathecal chemotherapy
* Tumors must be CD20+ on pathologic analysis
* Refractory or persistent disease allowed
* No complete obstruction of the CSF pathway within the ventricular system unless alleviated by external beam radiotherapy or systemic chemotherapy
* No obstructive hydrocephalus

PATIENT CHARACTERISTICS:

* Karnofsky performance status > 50%
* Must have an Ommaya reservoir
* Granulocyte count > 1,500/mm^3
* Platelet count > 50,000/mm^3
* Anticipated survival ≥ 1 month

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from toxicity of prior therapy
* Prior intrathecal methotrexate, cytarabine, or thiotepa for CNS lymphoma allowed
* Concurrent systemic chemotherapy for treatment of disease outside meninges allowed except for high-dose methotrexate, high-dose cytarabine, high-dose thiotepa, or investigational agents
* No history of whole-brain or craniospinal radiation < 1 week before study entry
* No history of intrathecal chemotherapy < 1 week before study entry
* No concurrent intrathecal chemotherapy

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2002-08; Primary Completion 2005-11 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Adverse events as a measure of safety of intrathecal administration of Rituximab | up to 5 years after completion of 5 week study treatment
Serum concentration of Rituximab | during 5 weeks of study treatment
Cerebrospinal Fluid (CSF) concentration of Rituximab | during 5 weeks of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: James L. Rubenstein, MD, PhD, Principal Investigator — University of California, San Francisco

REFERENCES:
- [Result] Rubenstein JL, Fridlyand J, Abrey L, Shen A, Karch J, Wang E, Issa S, Damon L, Prados M, McDermott M, O'Brien J, Haqq C, Shuman M. Phase I study of intraventricular administration of rituximab in patients with recurrent CNS and intraocular lymphoma. J Clin Oncol. 2007 Apr 10;25(11):1350-6. doi: 10.1200/JCO.2006.09.7311. Epub 2007 Feb 20. PMID 17312328